CLINICAL TRIAL: NCT05163197
Title: Transperineal Laser Ablation Treatment for Prostate Cancer Registry: a Retrospective and Multicenter Evaluation
Brief Title: Transperineal Laser Ablation Treatment (TPLA) for Prostate Cancer (PCa) Registry
Acronym: TPLAforPCa
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof.dr. H.P. Beerlage, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_458
Record Dates: First submitted 2021-10-28; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: Laser Ablation; Minimal invasive; Focal therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transperineal Laser Ablation of Prostate Cancer — Minimal invasive transperineal laser ablation treatment for prostate cancer
  Other Names: Soractelite treatment; Echolaser X4

SUMMARY:
Rationale: Transperineal laser ablation (TPLA) treatment for prostate cancer (PCa) is a minimal invasive focal therapy technique studied worldwide to determine its efficacy. In pilot studies it has shown to be a safe and feasible technique and it has potential to preserve continence and potency over current standard radical therapies. However, (long-term) treatment outcomes of TPLA for PCa remain largely unknown. The aim of this international retrospective registry is to collect and combine data on patients treated TPLA for PCa in order to provide data on safety, feasibility, functional and oncological outcomes.

Objective: To assess safety and feasibility of TPLA for PCa, to assess functional and oncological outcomes of TPLA for PCa and to determine baseline patient characteristics in a multicentre cohort.

Study design: This is an international, retrospective observational registry in which data is recorded of patients who have been treated with TPLA for PCa.

Study population: Male patients treated with TPLA for PCa. Main study parameters/endpoints: The primary endpoint of this registry is oncological outcomes of TPLA for PCa. Secondary endpoints are safety, feasibility and functional outcomes of TPLA for PCa.

ELIGIBILITY:
Inclusion Criteria:

* Male, histological-confirmed disease of localized prostate cancer, TPLA treatment for PCa is performed

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population comprises those patients that have been treated with TPLA for PCa.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Oncological control | 12 months
  Oncological control is defined as: a PSA <=2.0ng/mL than initial PSA and/or no residual tumor or other lesion suspicious for prostate cancer on magnetic resonance imaging and/or no gleason score upgrading on re-biopsy and/or no clinical up-staging of prostate cancer T-stage

SECONDARY OUTCOMES:
Continence rate | 12 months
  Continence is assessed by usage of number of pads per day, and 0-1 pad per day usage is defined as continent.
Potency rate | 12 months
  Potency is defined as erectile function sufficient for sexual intercourse, with or without medical aid
Urinary flow | 12 months
  Urinary flow is assessed by peak urinary flow (mL/s) and residual urine (mL). The higher the peak urinary flow and the lower the residual urine, the better the urinary flow.
PROM regarding voiding | 12 months
  International Prostate Symptom Score (IPSS) is used to determine functional outcome regarding voiding. IPSS is on a score of 0 to 35, and the higher the score the worse the outcome.
PROM regarding erectile function | 12 months
  International Index of Erectile Function (IIEF-5) is used to determine erectile function based on a validated questionnaire. IIEF-5 is on a scale of 5 to 25, and the higher the score the better the outcome.
Safety of TPLA for PCa | Up to 12 weeks
  Safety is defined as 10% or less CTCAE (version 5) grade 3 and no CTCAE grade 4 or 5
Feasibility of TPLA for PCa | Up to 4 weeks
  Feasibility is assessed by amount of machine failures perioperatively of TPLA and hospital duration (hours) directly after TPLA.

CONTACTS AND LOCATIONS:
Overall Officials: J. R. Oddens, MD, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Amsterdam University Medical Centers, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No